CLINICAL TRIAL: NCT02803866
Title: Assessing Parenting Self-efficacy Before and After Applying a Specific Training Program for Parents (CAP-PREM: Preterm Capacitation) During Hospitalization of Preterm Neonates
Brief Title: Training Parenting Self-efficacy in Parents of Hospitalized Preterm Neonates
Acronym: CAP-PREM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Manuel Sanchez Luna, Dr., Hospital General Universitario Gregorio Marañon
Other Study IDs: CCF-Padres 01
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Parenting; Preterm Infants; Training Support
Keywords: Parenting Self-efficacy; Parent training program; Perceived self-efficacy tool

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Parents of preterm newborns (25-32 weeks of gestation): Parents (mother or mother+father) of preterm newborns admitted at the Gregorio Marañón Hospital from birth, recruited during the first 10 days of preterm newborn hospitalization and receiving the training program CAP-PREM
  Interventions: Behavioral: Training program CAP-PREM

INTERVENTIONS:
Behavioral: Training program CAP-PREM — 1ºAfter recruitment parents will fill the PMP S-E tool and the psychological tests evaluating their stress and depression . 2º parents will receive the training program during 4 weeks. 3º: before hospital discharge parents will fill again the PMP S-E tool and the psychological test evaluating their depression and anxiety

SUMMARY:
In a hospital environment, initial parenting of a family with a preterm neonate will be very different than expected. This unusual and stressful situation may determine the self-confidence perceived by mothers and fathers in caring their baby and therefore could shape future interaction with him/her as well as neurodevelopmental and behavioral development of preterm infants.

24/7 neonatal units allow parents stay with their baby whenever they want but this free access nor guarantee neither encourage parenting self-efficacy if it isn't hand in hand with a specific training program for parents.

DETAILED DESCRIPTION:
Longitudinal, prospective, analytic cohort study of parents of preterm newborns who will receive a specific training program for caring their preterm newborns during hospitalization. Families will be recruited during the first 10 days of hospitalization. The PMP S-E (Perceived Maternal Parenting Self- Efficacy) tool developed by Barnes and Adamson-Macedo, will be used to measure self-efficacy in providing infant care by mother or both mother and father. The training program will be developed at bed side by nurses and neonatologist covering theoretical and practical sessions during the first 25 days of hospitalization.

Hypothesis principal: Parents of hospitalized preterm neonates will get better score after application of a specific training program (CAP-PREM).

Secondary hypothesis:

* There is a correlation between the level of stress and anxiety in parents at admission and discharge and the results of PMP S-E score after the CAP-PREM program
* To assess those selected demographic variables that can predict a better result in PMP S-E score after the CAP-PREM program

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants between 25 and 32 weeks of gestation,
* parents stay at the unit for at least 8 hours/day during training program
* fluent Spanish.
* parents age > 18 years
* No clinical instability, invasive mechanical ventilation, intraventricular hemorrhage >II or necrotizing enterocolitis .
* no congenital malformation nor chromosomal abnormalities

Exclusion criteria :

* No possibility of survival beyond the first week of life
* Admission less than 4 weeks
* No collaboration / lack of parental compliance
* wish of parents to leave the study

Ages: 10 Days to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Parents of hospitalized preterm neonates
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Perceive parental self-efficacy before and after CAP-PREM program | 4 weeks
  Training parents for caring their preterm newborn from the first days of hospitalization will give them the opportunity to be active parents and improve their perceive parenting

SECONDARY OUTCOMES:
Influence of parents' psychological state in acquiring self-efficacy | 4 weeks
  The emotional situation of parents during their preterm neonate hospitalization may interfere with their perceived parenting sel-efficacy
Explore which demographic data may predict the PMP S-E score | 4 weeks
  Gestational age, weeks of gestation,parity, first time of kangaroo care,

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Caballero, PhD, Principal Investigator — Gregorio Marañón Hospital
Locations (1):
- Sylvia Caballero, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes CR, Adamson-Macedo EN. Perceived Maternal Parenting Self-Efficacy (PMP S-E) tool: development and validation with mothers of hospitalized preterm neonates. J Adv Nurs. 2007 Dec;60(5):550-60. doi: 10.1111/j.1365-2648.2007.04445.x. PMID 17973719